CLINICAL TRIAL: NCT03573050
Title: Multiple Dose Crossover Comparative Bioavailability Study of a Transdermal Patch Formulation of Rivastigmine Compared With Exelon® Transdermal Patch With a Release Rate of 13.3 mg/24 Hours in Healthy Male Subjects With Preceding Adaptation Phase and Post-treatment Tapering Phase
Brief Title: Rivastigmine BA Trial With Multiple Application of Transdermal Patches, Adaptation and Tapering Phase
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Collaborators: SocraMetrics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1351riv18ct; 2018-000968-28 (EudraCT Number); C_30170_P1_16 (Other: Luye Pharma AG / Luye Supply AG)
Record Dates: First submitted 2018-05-22; First posted 2018-06-29 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Rivastigmine; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIV-TDS 13.3 mg/24 h (Test) (Experimental): 5 consecutive patch applications of Test (each patch to be applied for 24 hours)
  Interventions: Drug: RIV-TDS 13.3 mg/24 h
- Exelon® 13.3 mg/24 hours transdermal patch (Reference) (Active Comparator): 5 consecutive patch applications of Reference (each patch to be applied for 24 hours)
  Interventions: Drug: Exelon® 13.3 mg/24 hours transdermal patch

INTERVENTIONS:
Drug: RIV-TDS 13.3 mg/24 h — 5 consecutive transdermal patch applications, each with a nominal release rate of 13.3 mg/24 hours
  Arms: RIV-TDS 13.3 mg/24 h (Test)
Drug: Exelon® 13.3 mg/24 hours transdermal patch — 5 consecutive transdermal patch applications, each with a nominal release rate of 13.3 mg/24 hours
  Arms: Exelon® 13.3 mg/24 hours transdermal patch (Reference)

SUMMARY:
The present clinical trial will be conducted to compare the bioavailability of rivastigmine and assess bioequivalence at steady-state of the Test product RIV-TDS 13.3 mg/24 h and the marketed Reference product Exelon® 13.3 mg/24 hours transdermal patch after multiple patch application. Each of both treatments will last 5 days.

DETAILED DESCRIPTION:
This will be a single centre, open-label, randomised (order of treatments), balanced, 2-period, 2-sequence, cross-over trial with multiple applications of rivastigmine transdermal patches. There will be no wash-out, i.e. the first investigational patch application of the second study period will take place the day of the last investigational patch removal of the first study period (direct switch-over).

Prior to start of first treatment, there will be an adaptation phase with 4 consecutive applications of Exelon® 9.5 mg/24 hours transdermal patch over a period of 4 days (each patch will be applied for 24 hours). Following the removal of the last investigational patch in period II, there will be a post-treatment tapering phase with 2 consecutive applications of Exelon® 9.5 mg/24 hours transdermal patch over a period of 2 days (each patch will be applied for 24 hours).

Furthermore, during the adaptation phase, both study periods and the tapering phase, scopolamine transdermal patches will be applied as co-medication to attenuate effects of rivastigmine and reduce Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male
2. Ethnic origin: Caucasian
3. Age: 18 - 50 years, inclusive
4. Body-mass index2 (BMI): >=18.5 kg/m² and <= 30.0 kg/m²
5. Good state of health
6. Non-smoker or ex-smoker for at least 6 months
7. Written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

1. Existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredients (especially sick sinus syndrome or conduction defects such as sino-atrial block, atrio-ventricular block, arrhythmia, bradycardia)
2. Existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredients (especially predisposition to urinary obstruction and seizures or other conditions with difficulty in passing water owing to an impeded flow of urine (e.g. in diseases of the prostate))
3. Existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredients (especially active gastric or duodenal ulcers or predisposition to these conditions, pyloric stenosis, intestinal obstruction)
4. History of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders (e.g. cerebral sclerosis)
5. History of asthma or obstructive pulmonary disease
6. Glaucoma or any indications from case history that there might be raised intra-ocular pressure (e.g. pressure pain, blurred vision, glaucomatous halo)
7. Known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations or previous history of application site reactions suggestive of allergic contact dermatitis with rivastigmine or scopolamine patch
8. Subjects with severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
9. Body weight below 65 kg
10. Systolic blood pressure < 90 or ≥ 140 mmHg
11. Diastolic blood pressure < 60 or >90 mmHg
12. Heart rate < 60 bpm or > 90 bpm
13. QTc interval > 450 ms
14. Laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
15. ASAT > 20 % ULN, ALAT > 10 % ULN, bilirubin > 20% ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to of > 9 μmol/l ULN).
16. Positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test or anti-HCV-test
17. Presence or history of acute or chronic diseases especially of the skin, which could affect dermal absorption or metabolism, which may interfere with the bioavailability and /or the pharmacokinetics of scopolamine or rivastigmine patches based on assessment of the investigator
18. Skin abnormality (e.g. tattoo or scar) at the application site
19. Acute or chronic diseases which may interfere with the pharmacokinetics of scopolamine or rivastigmine patches
20. History of or current drug or alcohol dependence
21. Positive alcohol or drug test at screening examination
22. Regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol per day
23. Subjects who are on a diet which could affect the pharmacokinetics of the active ingredients
24. Regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
25. Blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the subject
26. Administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the subject
27. Regular treatment with any systemically available medication
28. Subjects practising top-performance sports (more than 4 x 2 h per week)
29. Subjects suspected or known not to follow instructions
30. Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial -

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
AUC0-tau,ss | from 0 to 24 hours following the 5th patch application
  Area under the plasma concentration vs. time curve at steady state for rivastigmine
Ctau,ss | from 0 to 24 hours following the 5th patch application
  (Trough) minimum plasma concentration at the end of the dosing interval at steady state for rivastigmine
Cmax,ss | from 0 to 24 hours following the 5th patch application
  Maximum plasma concentration within the dosing interval at steady state for rivastigmine

SECONDARY OUTCOMES:
Patch adhesion | from first investigational patch application until removal of the last investigational patch (approx. 10 days)
  one-sided lower 90% confidence limit of mean adherence percentage at the end of the dosing interval of the 5th patch
Skin irritation | from first investigational patch removal until last investigational patch removal (approx. 10 days)
  frequency of scores for quantification of skin irritation per treatment and time point
Adverse events | approximately 2 weeks, through study completion in case of follow-up
  descriptive evaluation of frequency and intensity, relationship to the IMP, action taken, outcome, seriousness, period and treatment

CONTACTS AND LOCATIONS:
Locations (1):
- SocraTec R&D GmbH, Clinical Pharmacology Unit, Erfurt, Thuringia, Germany

REFERENCES:
- [Derived] Morte A, Vaque A, Iniesta M, Schug B, Koch C, De la Torre R, Schurad B. Bioavailability Study of a Transdermal Patch Formulation of Rivastigmine Compared with Exelon in Healthy Subjects. Eur J Drug Metab Pharmacokinet. 2022 Jul;47(4):567-578. doi: 10.1007/s13318-022-00778-5. Epub 2022 Jun 13. PMID 35696054